CLINICAL TRIAL: NCT04050436
Title: A Randomized, Controlled, Open-Label, Phase 2 Study of Cemiplimab as a Single Agent and in Combination With RP1 in Patients With Advanced Cutaneous Squamous Cell Carcinoma
Brief Title: Study Evaluating Cemiplimab Alone and Combined With RP1 in Treating Advanced Squamous Skin Cancer
Acronym: CERPASS
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Replimune Inc. (Industry)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RPL-002-18
Record Dates: First submitted 2019-08-02; First posted 2019-08-08 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2025-01

CONDITIONS: Cutaneous Squamous Cell Carcinoma; Advanced Cutaneous Squamous Cell Carcinoma; Metastatic Cutaneous Squamous Cell Carcinoma
Keywords: Oncolytic Virus; Carcinoma; Carcinoma, Squamous Cell; Cemiplimab; Metastatic Cutaneous Squamous Cell Carcinoma; Oncolytic Immuno-gene therapy
MeSH Terms: conditions — Carcinoma; Carcinoma, Squamous Cell | interventions — cemiplimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cemiplimab in combination with RP1 (Experimental): Cemiplimab administered intravenously every 3 weeks in combination with RP1 administered as an intratumoral injection every 3 weeks
  Interventions: Drug: Cemiplimab; Biological: RP1
- Cemiplimab (Active Comparator): Cemiplimab administered intravenously as a single therapy every 3 weeks
  Interventions: Drug: Cemiplimab

INTERVENTIONS:
Drug: Cemiplimab — Cemiplimab administered intravenously
  Other Names: Libtayo
Biological: RP1 — RP1 administered intratumorally
  Other Names: Genetically modified herpes simplex type 1 virus
  Arms: Cemiplimab in combination with RP1

SUMMARY:
To estimate the clinical benefit of cemiplimab monotherapy versus cemiplimab in combination with RP1 for patients with locally advanced or metastatic CSCC, as assessed by overall response rate (ORR) and complete response rate (CRR) according to blinded independent review.

DETAILED DESCRIPTION:
RP1 is a selectively replication competent herpes simplex virus type 1(HSV-1). This is a Phase 1/2, open-label, multicenter repeat-dosing study of RP1 alone and in combination with nivolumab in patients with advanced malignancies, and contains both single agent dose escalation, dose expansion to include nivolumab, and the combination in multiple Phase 2 cohorts in individual tumor types.

ELIGIBILITY:
Key Inclusion Criteria:

* Histologically confirmed locally advanced or metastatic cutaneous squamous cell carcinoma
* Patients with locally advanced disease who are not suitable candidates for surgical or radiological treatment of lesions or have refused those treatments
* At least 1 lesion that is measurable and injectable by study criteria
* Eastern Cooperative Oncology Group (ECOG) performance status ≤1. Patients with ECOG PS 2 at baseline may be allowed to enroll if PS 2 status is only related to the CSCC disease under study
* Anticipated life expectancy >12 weeks
* All patients must consent to provide archived or newly obtained tumor material for central pathology review for confirmation of diagnosis of CSCC.

Key Exclusion Criteria:

* Prior treatment with an oncolytic therapy
* Patients with active significant herpetic infections or prior complications of HSV-1 infection (e.g. herpetic keratitis or encephalitis)
* Patients who require intermittent or chronic use of systemic (oral or intravenous) anti-virals with known anti-herpetic activity (e.g. acyclovir)
* Ongoing or recent (within 5 years) evidence of significant autoimmune disease that required treatment with systemic immunosuppressive treatments
* Prior treatment with an agent that blocks the PD-1/PD-L1 pathway.
* Prior treatment with other immune modulating agents other than as adjuvant or neoadjuvant therapy within 3 years.
* Untreated brain metastasis(es) that may be considered active.
* Acute or chronic active hepatitis B or known history of hepatitis B or hepatitis C or human immunodeficiency virus (HIV) infection
* History of ILD/pneumonitis within the last 5 years or a history of ILD/pneumonitis requiring treatment with systemic steroids.
* Any major or surgical procedure ≤ 28 days before randomization
* Administration of live vaccines ≤ 28 days before randomization

Note: Other protocol defined Inclusion/Exclusion criteria apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 231 (Actual)
Dates: Start 2019-10-08 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) according to blinded independent review | up to 5 years
Complete Response Rate (CRR) according to blinded independent review | up to 5 years

SECONDARY OUTCOMES:
Progression Free Survival (PFS) by blinded independent review. | up to 5 years
ORR/CRR by investigator assessment and blinded independent review | up to 5 years
ORR/CRR for patients with metastatic or locally advanced disease according to investigator review and blinded independent review | up to 5 years
ORR/CRR for patients who have and have not previously received systemic CSCC-directed therapy and blinded independent review | up to 5 years
Duration of Response (DOR) per investigator review and blinded independent review | up to 5 years
Progression-free Survival (PFS) per investigator review | up to 5 years
Overall Survival (OS) | up to 5 years
3-year survival | 3 years
Change in overall scores of patient-reported outcomes in European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30) | approximately 30 months
Evaluation of the safety and tolerability of cemiplimab alone and combined with RP1 as assessed via adverse events (AEs) | approximately 26 months

CONTACTS AND LOCATIONS:
Overall Officials: Moran Mishal, MD, Study Director — Lead Medical Monitor; Jeannie Hou, MD, Study Director — Secondary Medical Monitor
Locations (56):
- United States (14):
  - University of California San Diego, La Jolla, California
  - University of California Los Angeles, Los Angeles, California
  - Stanford University, Stanford, California
  - University of Colorado Cancer Center, Aurora, Colorado
  - University of Miami Health System, Miami, Florida
  - Orlando Health UF Health Cancer Center, Orlando, Florida
  - Moffitt McKinley Outpatient Center, Tampa, Florida
  - Winship Cancer Institute of Emory University, Atlanta, Georgia
  - John Theurer Cancer Center at Hackensack Univeristy Medical Center, Hackensack, New Jersey
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - University Of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Prisma Health Cancer Institute, Greenville, South Carolina
  - MD Anderson Cancer Center, Houston, Texas
- Australia (7):
  - Chris O'Brien Lifehouse, Camperdown, New South Wales
  - Cancer Care Wollongong Pty Limited, Wollongong, New South Wales
  - Tasman Oncology Research Ltd, Southport, Queensland
  - Monash Medical Centre, Clayton, Victoria
  - Peter MacCallum Cancer Centre, Melbourne, Victoria
  - The Alfred Hospital, Melbourne, Victoria
  - Sir Charles Gairdner Hospital, Nedlands, Western Australia
- Bulgaria (2):
  - Multiprofile Hospital for Active Treatment - Uni Hospital" OOD Department of Medical Oncology, Panagyurishte
  - "Complex Oncology Center - Plovdiv" EOOD Department of Medical Oncology and Cutaneous Cancer Diseases ", Plovdiv
- Sunnybrook Health Science Centre, Toronto, Ontario, Canada
- France (10):
  - CHU Besancon - Hopital Jean Minjoz, Besançon
  - CHU Dijon Hopital F. Mitterrand Service de Dermatologie - UMAC, Dijon
  - CHU de Grenoble - Hopital A Michallon, La Tronche
  - CHRU de Lille, Lille
  - Centre Léon Bérard, Lyon
  - Service de Dermatologie et Cancerologie Cutanee Hopital de la Timone, Marseille
  - CHU Nice - Hopital de l'Archet 2, Nice
  - Hospital Saint Louis, Paris
  - Hospices Civils de Lyon, Pierre-Bénite
  - Institut Gustave Roussy, Villejuif
- Germany (6):
  - Charite Universitatsmedizin Berlin, Berlin
  - Universitatsklinikum Essen, Essen
  - Universitätsklinikum Eppendorf, Hamburg
  - Universitatsklinikum Heidelberg: National Centre for Tumour Diseases (NCT), Heidelberg
  - University Hospital Munchen (LMU), München
  - Universitatsklinikum Tubingen Zentrum fur Dermatoonkologie, Tübingen
- Greece (4):
  - Hippocratio General Hospital of Athens, Athens
  - Attiko University Hospital, Athens
  - Andreas Syggros Hospital, Athens
  - General Hospital of Athens "Laiko", 1st Department of Medicine, University of Athens Medical School, Athens
- Istituto Tumori "Giovanni Paolo II" IRCCS, Bari, Italy
- Poland (4):
  - Uniwersyteckie Centrum Kliniczne; Centrum Leczenia Czerniaka w Gdańsku, Gdansk
  - Narodowy Instytut Onkologii; Panstwowy Instytut Badawczy Oddzial w Krakowie, Krakow
  - Narodowy Instytut Onkologii; Panstwowy Instytut Badawczy, Warsaw
  - Klinika Dermatologii, Wenerologii i Alergologii, USK im J. Mikulicza-Radeckiego we Wroclawiu, Wroclaw
- Spain (7):
  - Hospital Clinic Barcelona, Barcelona
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario Fundación Jiménez Díaz, Madrid
  - Hospital Universitario Virgen de la Arrixaca, Murcia
  - Clinica Universitaria de Navarra, Pamplona
  - Hospital General Universitario De Valencia, Valencia

IPD SHARING:
Plan to Share IPD: No